CLINICAL TRIAL: NCT03169361
Title: NINLARO Capsules Drug Use-Results Survey (All-Case Surveillance) "Relapsed/Refractory Multiple Myeloma"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16025; JapicCTI-173592 (Registry Identifier: Japic-CTI)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ixazomib 4 mg: The usual adult dosage for oral administration is 4 mg as ixazomib, in the fasting state, once a day, once a week for 3 weeks (Days 1, 8, and 15), with a 13-day washout period (Days 16 through 28). This 4-week cycle will be repeated for 6 cycles. The dose may be reduced appropriately according to the patient's condition. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: NINLARO capsules; MLN9708

SUMMARY:
The purpose of this study is to evaluate the safety of NINLARO in participants with relapsed/refractory multiple myeloma in daily clinical practice.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib (NINLARO). Ixazomib is being tested to treat people who have relapsed/refractory multiple myeloma. This study will look at the safety of NINLARO in participants with relapsed/refractory multiple myeloma in daily clinical practice.

The study will enroll approximately 480 patients.

• Ixazomib 4 mg

This multi-center trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been confirmed as administration of the drug.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all participants with a diagnosis of multiple myeloma and received their first dose of NINLARO/lenalidomide, and dexamethasone.
Sampling Method: Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60204db2bf003ab49567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 316 investigative sites in Japan, from 24 May 2017 to 8 March 2022.
Pre-assignment Details: Participants with a historical diagnosis of relapsed/refractory multiple myeloma were enrolled. Participants received ixazomib as part of a routine medical care.
Groups:
- Ixazomib 4 mg: The usual adult dosage for oral administration was 4 mg as ixazomib, in the fasting state, once a day, once a week for 3 weeks (Days 1, 8, and 15), with a 13-day washout period (Days 16 through 28). This 4-week cycle was repeated for 6 cycles. The dose might be reduced appropriately according to the patient's condition. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Ixazomib 4 mg
Started | 774
Completed | 742
Not Completed | 32
Not completed — Protocol Violation | 32

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Ixazomib 4 mg
Number analyzed (Participants) | 742
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391
  Male | 351
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 742
Duration of Diagnosis of Relapsed/Refractory Multiple Myeloma [Mean (Standard Deviation); unit: Years] — Mean duration between the first diagnosis of relapsed/refractory multiple myeloma and the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 739
    (all) | 4.49 (3.902)
Number of Participants with Relapsed/Refractory Multiple Myeloma [Count of Participants; unit: Participants] | 742
International Staging System [Count of Participants; unit: Participants] — International Staging System is a staging system for cancer progression. Stages are classified by Stage I to Stage III. Stage I: Serum beta2-microglobulin <3.5 mg/L and albumin ≥3.5 g/dL; Stage II: Neither Stage I or III, meaning that either: beta2-microglobulin level ≥3.5 and <5.5 mg/L (with any albumin level), OR albumin <3.5 g/dL with beta2-microglobulin <3.5 mg/L; Stage III: Serum beta2-microglobulin ≥5.5 mg/L. Normal serum beta2-microglobulin: <3.0 mg/L; normal albumin: 3.5-5.0 g/dL. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 740
    Stage I | 140
    Stage II | 260
    Stage III | 290
    Missing | 50
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status assess participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50 percent [%] of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead.
  Participants
    Scale = 0 | 240
    Scale = 1 | 294
    Scale = 2 | 112
    Scale = 3 | 81
    Scale = 4 | 15
Healthcare Category [Count of Participants; unit: Participants]
  Outpatient | 436
  Inpatient | 306
Hepatic Impairment [Count of Participants; unit: Participants]
  Had No Hepatic Impairment | 696
  Had Hepatic Impairment | 46
Renal Impairment [Count of Participants; unit: Participants]
  Had No Renal Impairment | 448
  Had Renal Impairment | 294
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 741
    Had No Medical Complications | 307
    Had Medical Complications | 434
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 741
    Had No Medical History | 475
    Had Medical History | 259
    Unknown | 7
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 715
    (all) | 156.2 (10.01)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 709
    (all) | 54.10 (11.764)
Body Surface Area [Mean (Standard Deviation); unit: Square Meter] — Population: The number analyzed is the number of participants with data available for analysis.
  Square Meter
    number analyzed (Participants) | 705
    (all) | 1.53 (0.204)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 24 Week (From start of administration to the end of 6 cycles)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4 mg
Number analyzed (Participants) | 742
Participants | 642

2. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions (ADRs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction (ADR) refers to AE related to administered drug.
Time Frame: Up to 24 Week (From start of administration to the end of 6 cycles)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4 mg
Number analyzed (Participants) | 742
Participants | 573

ADVERSE EVENTS:
Time Frame: Up to 24 Week (From start of administration to the end of 6 cycles)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded. The data reported are only serious and the other (not including serious) ADRs by events because only serious and the other ADRs were planned to be collected and assessed in this study. Seriousness of AEs by events was out of the scope for the data collection plan.
Arm/Group | Ixazomib 4 mg
All-Cause Mortality (participants affected / at risk) | 11/742
Serious Adverse Events (participants affected / at risk) | 193/742
Other Adverse Events (participants affected / at risk) | 515/742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg (N=742)
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 5
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 22
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia haemophilus (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Septic shock (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Candida sepsis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Intervertebral discitis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 3
Herpes zoster disseminated (Infections and infestations) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 73
Dehydration (Metabolism and nutrition disorders) | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 7
Altered state of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 7
Thalamus haemorrhage (Nervous system disorders) | 1
Autonomic neuropathy (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 2
Atrioventricular block second degree (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Stress cardiomyopathy (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 2
Hypovolaemic shock (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 44
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Pancreatitis acute (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 17
Tongue haemorrhage (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 6
Prerenal failure (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Malaise (General disorders) | 4
Oedema (General disorders) | 1
Pyrexia (General disorders) | 3
Blood lactate dehydrogenase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 9
C-reactive protein increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg (N=742)
Thrombocytopenia (Blood and lymphatic system disorders) | 313
Neuropathy peripheral (Nervous system disorders) | 45
Diarrhoea (Gastrointestinal disorders) | 178
Nausea (Gastrointestinal disorders) | 82
Vomiting (Gastrointestinal disorders) | 52
Rash (Skin and subcutaneous tissue disorders) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT03169361/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT03169361/SAP_001.pdf